CLINICAL TRIAL: NCT00966992
Title: Randomized Phase II Study of Zoledronic Acid vs Observation on Bone Mineral Density and Incidence of Micrometastasis in Women Undergoing Pelvic Radiation for Cervical Cancer
Brief Title: Study of Zoledronic Acid Versus Observation on Bone Mineral Density and Incidence of Micrometastasis in Women Undergoing Pelvic Radiation for Cervical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-0811
Record Dates: First submitted 2009-08-18; First posted 2009-08-27 (Estimated); Results first posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-08

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Uterine Cervical Cancer; Cancer of Cervix; Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (No Zometa) (No Intervention): Women will complete their standard chemoradiation treatment protocol and end of treatment PET scan at about 3 months from completion of radiation. All interventions on this arm are standard of care.
- Arm 2 (Zometa) (Experimental): Women will complete their standard chemoradiation treatment protocol and end of treatment PET scan at about 3 months from completion of radiation. Women randomized to zoledronic acid will receive 4 mg intravenously (IV) with their first dose chemotherapy and 3, 6 and 9 months after completion of radiation (total of 4 doses) along with scheduled follow-up dual-energy X-ray absorptiometry (DEXA) and biomarker studies.
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid
  Other Names: Zometa
  Arms: Arm 2 (Zometa)

SUMMARY:
The treatment of cervical cancer with chemotherapy and radiation will make women post menopausal (no estrogen from the ovaries), if a woman is not already in menopause. Estrogen plays a key role in maintaining bone health. Therefore, these women are at higher risk of getting osteoporosis (decrease minerals in the bone) and bone fractures. The overall purpose of this research is to look at the effects of zoledronic acid (Zometa) on preventing bone loss. Studies have also shown that zoledronic acid may prevent metastasis to the bone which can occur in women with cervical cancer. Zometa is investigational (not approved by the Food and Drug Administration (FDA)) in this study to prevent metastasis to the bone in women with cervical cancer. Therefore, the goal of this study is to also look at the effects of zoledronic acid (Zometa) on circulating tumor cells in the bone marrow and blood. This study is being done to find a way to prevent bone loss and metastasis to the bone in women undergoing chemotherapy and radiation for cervical cancer. An additional component of the study is to assess the importance of stress on immune markers in blood during standard treatment.

DETAILED DESCRIPTION:
OBJECTIVES

* To determine the incidence of disseminated tumor cells (DTCs) in bone marrow and circulating tumor cells (CTCs) in the blood of women with cervical cancer at diagnosis and 3 to 9 months after chemotherapy and pelvic radiation with and without Zometa.
* To determine the change in biochemical markers of bone turnover from diagnosis to 9 months after radiation in women receiving chemoradiation for cervical cancer with and without Zometa.
* To determine change in bone mineral density from diagnosis to 9 month after chemoradiation with and without Zometa.
* To determine if depressed and anxious mood are associated with greater impairment of adaptive immunity (ratio of Th1/Th2) and higher levels of angiogenesis (VEGF) in peripheral blood of cervical cancer patients.
* To examine the relationship of standardized uptake values (SUV)Max and metabolic heterogeneity in the primary tumor and evidence of persistent/recurrent disease on the 3 and 9 month Fludeoxyglucose (FDG)-Positron Emission Tomography (PET) scans with DTCs and CTCs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous, adenosquamous or adenocarcinoma International Federation of Gynecology and Obstetrics (FIGO) Stage IB-IVA of the uterine cervix undergoing initial radiation and cisplatin based chemotherapy for primary treatment.
* Gynecologic Oncology Group performance status of 0, 1, or 2.
* Patients with ureteral obstruction must undergo stent placement or nephrostomy tube placement prior to study entry.
* Age >= 18 years.
* Patients must have signed informed consent.
* Patients must have adequate:

  * Bone marrow function: absolute neutrophil count (ANC) greater than or equal to 1,500/ul, equivalent to Common Toxicity Criteria (CTCAE) grade 1. Platelets greater than or equal to 100,000/ul.
  * Renal function: creatinine less than or equal to 1.5 x institutional upper limit normal (ULN). If creatinine is greater than 1.5 x ULN, creatinine clearance must be greater than 60 ml/min.
  * Hepatic function: bilirubin less than or equal to 1.5 x ULN. AST and alkaline phosphatase less than or equal to 2.5 x ULN.
  * Neurologic function: neuropathy (sensory and motor) less than or equal to CTCAE grade 1.
  * Coagulation: prothrombin time (PT) such that the international normalized ratio (INR) is < 1.5 (INR may be between 2 and 3 if a patient is on stable dose of therapeutic warfarin) and a PTT < 1.2 times control.

Exclusion Criteria:

* Evidence of sepsis or severe infection.
* Previous or current treatment for osteoporosis. Patients with denovo osteoporosis are also excluded.
* Evidence of bone metastasis.
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), or exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g., extraction, implants).
* Patients with history of other invasive malignancy (treatment within the last 5 years) other than non-melanoma skin cancer.
* Patients with known hypersensitivity to Zometa or other bisphosphonates.
* Patients who are pregnant or breast feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry Grigsby, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 08/12/2009 and closed to participant enrollment on 08/31/2010.
Groups:
- Arm 2 (Zometa): Women will complete their standard chemoradiation treatment protocol and end of treatment PET scan at about 3 months from completion of radiation. Women randomized to zoledronic acid will receive 4 mg intravenously (IV) with their first dose chemotherapy and 3, 6 and 9 months after completion of radiation (total of 4 doses) along with scheduled follow-up dual-energy X-ray absorptiometry (DEXA) and biomarker studies.
  Zoledronic acid
Period: Overall Study
Arm/Group | Arm 1 (No Zometa) | Arm 2 (Zometa)
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (No Zometa) | Arm 2 (Zometa) | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 1 |  | 1
Gender [Number; unit: participants]
  Female | 3 |  | 3
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Circulating Tumor Cells (CTCs)
Time Frame: At time of diagnosis, 3 months after completion of treatment, and 9 months after completion of treatment
Population: This outcome measure could not be analyzed as there were no participants enrolled in the zometa arm and the outcome measure required comparing results from the no zometa arm to the zometa arm.
Arm/Group | Arm 1 (No Zometa) | Arm 2 (Zometa)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Incidence of Disseminated Tumor Cells in Bone Marrow
Time Frame: At time of diagnosis, 3 months after completion of treatment, and 9 months after completion of treatment
Population: as for outcome 1
Arm/Group | Arm 1 (No Zometa) | Arm 2 (Zometa)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Bone Mineral Density
Time Frame: At the time of diagnosis and 9 months after completion of treatment
Population: as for outcome 1
Arm/Group | Arm 1 (No Zometa) | Arm 2 (Zometa)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Biochemical Markers of Bone Turnover
Time Frame: At the time of diagnosis and 9 months after completion of treatment
Population: as for outcome 1
Arm/Group | Arm 1 (No Zometa) | Arm 2 (Zometa)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: If Depressed and Anxious Moods Are Associated With Greater Impairment of Adaptive Immunity and Higher Levels of Angiogenesis in Peripheral Blood
Time Frame: At diagnosis, 6 months after completion of treatment, and 9 months after completion of treatment
Population: as for outcome 1
Arm/Group | Arm 1 (No Zometa) | Arm 2 (Zometa)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Relationship of SUVmax and Metabolic Heterogeneity in the Primary Tumor and Evidence of Persistent/Recurrent Disease
Time Frame: 3 months after completion of treatment and 9 months after completion of treatment
Population: as for outcome 1
Arm/Group | Arm 1 (No Zometa) | Arm 2 (Zometa)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1 (No Zometa) | Arm 2 (Zometa)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (No Zometa) (N=3) | Arm 2 (Zometa) (N=0)
Hypertension (Vascular disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Hemoglobin (Investigations) | 1 | 0
Leukocytes (WBC) (Investigations) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Pelvis pain (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes